CLINICAL TRIAL: NCT04424680
Title: Evaluating the Efficacy of an Advanced Care Planning Program for Health Decisions in Patients With Advanced Heart Failure
Brief Title: Efficacy of an Advanced Care Planning Program in Advanced Heart FAilure
Acronym: EACPAHFA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Universitario Fundación Alcorcón (Other)
Responsible Party: Principal Investigator, Benjamín Herreros Ruiz Valdepeñas, Principal Investigator; Internal Medicine Unit, Hospital Universitario Fundación Alcorcón
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HUFAlcoron
Record Dates: First submitted 2020-05-29; First posted 2020-06-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Intervention Model Description: Once patients have been included in the study, the assignment process will be carried out by random sampling to the study groups. In the First Group (control group), patients will be followed in HF outpatients units according to the usual established protocol. In the Second Group (intervention group), patients will participate in the ACP program. Treatment for HF will be the same in both groups. The research team has developed the ACP program based on the published bibliography on ACP and advanced HF. The four hospitals mentioned will start recruiting at the beginning of the study. The principal investigator will be responsible for interrupting recruitment once the sample size has been reached.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Patients will be followed in heart failure outpatients units according to the usual established protocol. In the first visit, patients from both control and intervention groups will complete the questionnaires with the help of researchers. After one year of follow-up, the questionnaires will be submitted again to all patients and three new questionnaires will be proposed.
  Treatment for heart failure will be the same in both groups.
- Intervention (Experimental): Patients will participate in the Advanced Care Planning Program. In the first visit, patients from both control and intervention groups will complete the questionnaires with the help of researchers. After one year of follow-up, the questionnaires will be submitted again to all patients and three new questionnaires will be proposed.
  Treatment for heart failure will be the same in both groups.
  Interventions: Behavioral: Advanced Care Planning program of health decisions

INTERVENTIONS:
Behavioral: Advanced Care Planning program of health decisions — Application of an Advanced Care Planning program program for decision-making in patients with advanced Heart Failure, in comparison to usual follow up and care.
  Arms: Intervention

SUMMARY:
An "Advanced Planning Program of Health Decisions" (APPHD) is a process of reflection and relationship between the patient, their relatives and health professionals. It is based on respect for patient's autonomy, to engage patients in making decisions about their disease so that the process is shared between the medical team, the patient and their relatives. Until now, it has not been measured whether the APPHD is effective and, therefore, really fulfills its purpose

DETAILED DESCRIPTION:
BACKGROUND: An Advanced Care Planning (ACP) program of health decisions is the result of a process of reflection and relationship-building between the patient, their relatives and health professionals. It is based on respect for patients' autonomy, involving them in making decisions about their disease in a way that is shared between the medical team, the patient and their relatives. Up until now, the efficacy of an ACP has not been measured in the existing literature, and therefore it is unknown if these programs reach their goal. OBJETIVES: The main objective of our study is to evaluate the efficacy of an ACP program for decision-making in patients with advanced heart failure (HF) in comparison to usual follow up and care. This objective will be evaluated by the Patient Activation Measure test, which measures the participation and self-management of the patient in decision-making. Secondary objectives: to evaluate the effect of the program on quality of life, to know if the patients wishes expressed through the ACP program are fulfilled, to measure the impact of the program on patients' caregivers, to determine the satisfaction of patients included in the program and to evaluate the effect on quality of death. METHODS: randomized multicentre clinical trial at four hospitals in Madrid. Once they are included in the study, patients' allocation to groups (control vs intervention) will be made by alternative sampling. ACP will be applied to the intervention group, whereas in the Control Group usual follow-up will be carried out in HF units. All patients will fulfil questionnaires and tests related to the objectives of the study again after a 12-month follow-up period in order to gauge the effect of ACP in patients with advanced HF.

ELIGIBILITY:
Inclusion Criteria:

* Patients with HF defined by Framingham diagnostic criteria.
* Stage C or D of the ACCF / AHA classification.
* Full capacity to decide.
* Signing of informed consent.

Exclusion Criteria:

* Cognitive impairment, measured by Mini-Mental Status Examination (< 27).
* Presence of another disease other than HF that may severely affect the quality of life: stroke with significant residual deficit, end-stage renal failure, Child C cirrhosis, extreme obesity, haemoglobin <8 g / dl, advanced peripheral artery disease (stage III-IV), severe thyroid or adrenal disease, neoplastic with estimated survival of less than 2 years.
* Patients who do not sign the informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 140 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-03-31 (Estimated); Study Completion 2023-01-01 (Estimated)

PRIMARY OUTCOMES:
To evaluate the efficacy of an Advanced Care Planning program for decision-making in patients with advanced Heart Failure in comparison to usual follow up and care: questionnaire | 24 months
  This objective will be evaluated by the PAM (Patient Activation Measure) test, which measures the participation and self-management of the patient in decision making. PAM measures the activation (participation and self-management) of the patient in decision-making. It evaluates the knowledge, skills and confidence of patients' self-management classifying patients in levels of self-management activation. Level 1: They do not feel responsible for their own health and care. (Score 47.0 or lower); Level 2: They may lack basic understanding about their condition, treatment options, and / or self-care. (47.1 to 55.1); Level 3: They know the basic facts of their illness and treatments. (55.2 to 67); Level 4: They have made most of the decisions, but they may have difficulties in maintaining behaviours over time or in stressful situations (67.1 or higher).

SECONDARY OUTCOMES:
To evaluate the effect of the ACP program on quality of life: questionnaire | 24 months
  This objective will be evaluated by the LWHFQ Questionnaire (Minnesota Living with Heart Failure Questionnaire), which measures the quality of life in patients with HF. Scoring range: 0 to 105 points: The higher the score obtained, the poorer the quality of life of patients. Questions refer to signs and symptoms of the disease, social relationships, physical, sexual activity, work and emotions. It is self-administered, with Likert response options, ranging from 0 (quality of life not affected) to 5 (maximum impact on quality of life). The global score is obtained by adding the 21 items scores (range: 0-105); the highest value corresponds to the worst quality of life. It assesses the impact of chronic heart failure in two dimensions: the physical dimension based on eight items (range: 0-40) and the emotional dimension consisting of five items (range: 0-25).
To know if the patients wishes expressed through the ACP program are fulfilled | 24 months
  This objective will be evaluated by a Checklist to test the fulfilment of planned patient's wishes.
To determine the level of satisfaction with the ACP program of patients included in the program. | 24 months
  This objective will be evaluated by a Satisfaction test Created "ad hoc". It aims to assess the level of satisfaction with the program. Its outcome will help improve the future implementation of the program.
  Satisfaction test. Answer YES or NO
  * Did you understand what the Program was about?
  * Do you feel you received enough information, orally or in writing, for your understanding?
  * Did you feel that you could easily access the doctors responsible for the program to answer your questions?
  * Do you think that the doctors responsible for the program have the necessary skills and knowledge?
  * Did you understand without difficulty what these professionals communicated in each interview?
  * Has the program met your expectations and needs?
  * Did you find it easy to get to the office and / or day hospital?
To evaluate the effect on quality of death: questionnaire | 24 months
  This objective will be evaluated by the Dying and Death quality questionnaire (QODD). This questionnaire measures the quality of the dying process.
  Quality of Dying and Death - 17-Item Version: Each item includes a filter question reporting what actually occurred during the final period of the decedent's life, followed by a rating of what occurred. The first 10 filter questions ask the frequency of occurrence and use the following response options: 0: none of the time; 1: a little bit of the time ; 2: some of the time; 3: a good bit of the time; 4: most of the time; 5: all of the time. The last 7 filter questions ask whether the event occurred and are answered with a yes/no response. After each filter question, the respondent rates the decedent's experience, using the following scale: 0 = terrible experience…10 = almost perfect experience.
To measure the impact of the ACP program on patients' caregivers | 24 months
  This objective will be evaluated by the Zarit questionnaire about caregiver's burden.
  Zarit questionnaire about caregiver's burden. This interview measures caregivers' degree of subjective overload in relation to chronic patients. It consists of 22 items that collect caregivers' feelings. Each feeling scores on a frequency gradient that ranges from 1 (never) to 5 (almost always). Interpretation:
  * or <45 points: no overload
  * 47 to 55 points: slight overload
  * or> 55 points: intense overload

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario Fundación Alcorcón, Alcorcón, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
The databases to be managed will be anonymous
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 12 months
Access Criteria: Study investigators

REFERENCES:
- [Result] Perez M, Herreros B, Martin MD, Molina J, Kanouzi J, Velasco M. Do Spanish Hospital Professionals Educate Their Patients About Advance Directives? : A Descriptive Study in a University Hospital in Madrid, Spain. J Bioeth Inq. 2016 Jun;13(2):295-303. doi: 10.1007/s11673-016-9703-7. Epub 2016 Jan 21. PMID 26797513
- [Result] Perez M, Herreros B, Martin MD, Molina J, Guijarro C, Velasco M. [Changes in knowledge and carrying out the advance directives of patients admitted to internal medicine]. Rev Calid Asist. 2013 Sep-Oct;28(5):307-12. doi: 10.1016/j.cali.2013.03.008. Epub 2013 Sep 7. Spanish. PMID 24021533
- [Result] Molina J, Perez M, Herreros B, Martin MD, Velasco M. [Knowledge and attitude regarding previous instructions for the patients of a public hospital of Madrid]. Rev Clin Esp. 2011 Oct;211(9):450-4. doi: 10.1016/j.rce.2011.06.007. Epub 2011 Aug 2. Spanish. PMID 21813119
- [Result] Miles SH, Koepp R, Weber EP. Advance end-of-life treatment planning. A research review. Arch Intern Med. 1996 May 27;156(10):1062-8. PMID 8638992
- [Result] Gomez-Batiste X, Martinez-Munoz M, Blay C, Amblas J, Vila L, Costa X, Espaulella J, Villanueva A, Oller R, Martori JC, Constante C. Utility of the NECPAL CCOMS-ICO(c) tool and the Surprise Question as screening tools for early palliative care and to predict mortality in patients with advanced chronic conditions: A cohort study. Palliat Med. 2017 Sep;31(8):754-763. doi: 10.1177/0269216316676647. Epub 2016 Nov 4. PMID 27815556
- [Derived] Sanchez B, Guijarro C, Velasco M, Vicente MJ, Galan M, Herreros B. Evaluating the efficacy of an Advanced Care Planning Program for Health Decisions in patients with advanced heart failure: protocol for a Randomized Clinical Trial. BMC Cardiovasc Disord. 2020 Oct 21;20(1):456. doi: 10.1186/s12872-020-01738-0. PMID 33087061